CLINICAL TRIAL: NCT03400293
Title: RISE: Real World Insights of People Living With HIV Shared Through Electronic Devices
Brief Title: Real-world Insights of People With Human Immunodeficiency Virus (HIV) Infection
Acronym: RISE
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: Evidera (Industry); mProve (Unknown)
Responsible Party: Sponsor
Other Study IDs: 208141
Record Dates: First submitted 2018-01-10; First posted 2018-01-17 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: HIV Infections
Keywords: Human Immunodeficiency virus; Health Related Quality of Life; Functional Assessment of HIV Infection; Mobile app
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects living with HIV: Subjects living with HIV will be recruited via digital advertising. These subjects will participate in completing various PRO instruments and targeted questions.
  Interventions: Other: Functional Assessment of HIV Infection; Other: Patient Satisfaction Questionnaire; Other: Symptom Distress Module; Other: Patient Health Questionnaire; Other: Internalized Stigma of AIDS Tool; Other: Medication adherence visual analogue scale

INTERVENTIONS:
Other: Functional Assessment of HIV Infection — Functional Assessment of HIV Infection will be used to assess HRQoL of subjects. This will include 47 items.
Other: Patient Satisfaction Questionnaire — Patient Satisfaction Questionnaire will be used to assess burden and HRQoL in subjects. This will include 18 items.
Other: Symptom Distress Module — Symptom Distress Module will be used to assess burden and HRQoL in subjects. This will include 20 items.
Other: Patient Health Questionnaire — Patient Health Questionnaire will be used to assess burden and HRQoL in subjects. This will include 2 items.
Other: Internalized Stigma of AIDS Tool — Internalized Stigma of AIDS Tool will be used to assess burden and HRQoL in subjects. This will include 10 items.
Other: Medication adherence visual analogue scale — Medication adherence visual analogue scale will be used to assess burden and HRQoL in subjects. This will include 1 item.

SUMMARY:
This study is designed to identify the burden associated with HIV and its treatment, and assess their health-related quality of life (HRQoL) by measuring key HRQoL domains, including satisfaction with treatment and care, and internalised stigma (ISAT). The study will also explore data for various important subpopulations such as subjects who are virally suppressed; who we anticipate will be the majority of study subjects. The study design is an observational, cross sectional study employing subjects' own mobile phone devices for data entry.

ELIGIBILITY:
Inclusion Criteria:

* >= 21 years old
* Language:Read and Understand English / Spanish
* Positive diagnosis of HIV infection by a healthcare provider (self-reported)
* Possesses a smartphone that has internet access

Exclusion Criteria:

* Not Applicable

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PLHIV will be recruited advertising in digital media. The study plan is to collect a complete set of data from 3000 PLHIV during a 90-180 day period in the US.
Sampling Method: Non-Probability Sample
Enrollment: 1184 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-07-07 (Actual); Study Completion 2018-07-07 (Actual)

PRIMARY OUTCOMES:
Percentage of virally suppressed PLHIV reporting different HRQoL scores | Up to 1 Week
  Evaluation of HRQoL will be conducted using scores achieved by Functional Assessment of HIV Infection (FAHI). QoL assessment will include physical well-being, social well-being, emotional well-being, functional and global well-being, and cognitive functioning

SECONDARY OUTCOMES:
Percentage of virally suppressed PLHIV reporting different satisfaction with care scores | Up to 1 Week
  Evaluation of burden will include stigma, stigma, depression, and work productivity. The descriptive analysis will be assessed using Patient Satisfaction Questionnaire (PSQ)-18, Patient Health Questionnaire (PHQ)-2, and ISAT scores
Percent difference in HRQoL scores among subject subgroups | Up to 1 Week
  Subject subgroups are defined in terms of the following socio-demographic, clinical, and biomedical factors: a. Age: older versus. younger (i.e., < 50 years old and over 50 years old) b. Gender (men / women / transgender) c. Race / ethnicity d. Sexual orientation (straight / gay / bisexual) e. Level of income f. Type of Insurance g. Apple (iPhone operating system) versus Android users h. Treatment regimen (e.g., number of pills per day, frequency of medication, single treatment regimen (STR) versus multiple treatment regimen (MTR) i. Diagnosis time / stage at which diagnosis was received (i.e. prompt vs. late diagnosis, time since diagnosis) j. Absence or presence (and number) of comorbidities k. Severity of symptoms (as assessed by the Symptom Distress Module patient reported outcome (PRO) instrument) l. Achievement of viral suppression.
Percentage of subjects reporting different HRQoL scores and relationship with satisfaction with care | Up to 1 Week
  Statistical correlation of reported QoL scores (FAHI) and satisfaction with care scores (PHQ-18) will be analyzed.
Percentage of subjects reporting diffferent HRQoL and medication adherence | Up to 1 Week
  Statistical correlation between QoL scores (FAHI) and adherence scores (adherence VAS) will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Arlington, Virginia, United States